CLINICAL TRIAL: NCT05420454
Title: A Prospective, Open-label Study to Evaluate Injectable Albumin-bound Paclitaxel Versus Docetaxel for the Neoadjuvant Treatment of Breast Cancer
Brief Title: A Study for the Neoadjuvant Treatment of Breast Cancer
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0055
Record Dates: First submitted 2022-06-12; First posted 2022-06-15 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Breast Cancer
Keywords: breast cancer; neoadjuvant therapy; Docetaxel; albumin-bound paclitaxel; TCbHP; nPCbHP; ddEC-wnP; EC-T
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Carboplatin; Trastuzumab; pertuzumab; Taxes; Epirubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- TCbHP (Active Comparator): HER2-positive breast cancer
  Interventions: Drug: Docetaxel; Drug: Carboplatin; Drug: Trastuzumab; Drug: Pertuzumab
- nPCbHP (Experimental): HER2-positive breast cancer
  Interventions: Drug: Carboplatin; Drug: Trastuzumab; Drug: Pertuzumab; Drug: Nab paclitaxel
- EC-T (Active Comparator): Luminal breast cancer (HER2-, LN+), and triple negative breast cancer
  Interventions: Drug: Epirubicin; Drug: Cyclophosphamide; Drug: Docetaxel
- ddEC-wnP (Experimental): Luminal breast cancer (HER2-, LN+), and triple negative breast cancer
  Interventions: Drug: Epirubicin; Drug: Cyclophosphamide; Drug: Nab paclitaxel

INTERVENTIONS:
Drug: Docetaxel — 75 mg/m2, d1, q3w,6 cycles
  Arms: TCbHP
Drug: Carboplatin — AUC 6, d1, q3w ,6 cycles
  Arms: TCbHP; nPCbHP
Drug: Trastuzumab — starting dose 8 mg/kg, maintenance dose 6 mg/kg, d1, q3w ,6 cycles
  Arms: TCbHP; nPCbHP
Drug: Pertuzumab — starting dose of 840 mg, maintenance dose of 420 mg, d1, q3w,6 cycles
  Arms: TCbHP; nPCbHP
Drug: Nab paclitaxel — 220 mg/m2, d1, q3w,6 cycles
  Arms: nPCbHP
Drug: Epirubicin — 90 mg/m2,d1, q3w × 4 cycles,followed by docetaxel
  Arms: EC-T
Drug: Cyclophosphamide — 600 mg/m2, d1, q3w ,4 cycles,followed by docetaxel
  Arms: EC-T
Drug: Docetaxel — 100 mg/m2, d1, q3w × 4 cycles
  Arms: EC-T
Drug: Epirubicin — 90 mg/m2,d1, q2w × 4 cycles,followed by nab-paclitaxel
  Arms: ddEC-wnP
Drug: Cyclophosphamide — 600 mg/m2, d1, q2w × 4 cycles followed by nab-paclitaxel
  Arms: ddEC-wnP
Drug: Nab paclitaxel — 125 mg/m2, d1,8,15, q3w× 4 cycles
  Arms: ddEC-wnP

SUMMARY:
Due to the unique advantages of albumin-bound paclitaxel, several studies in China and abroad have tried to use albumin-bound paclitaxel for neoadjuvant treatment of breast cancer up to now. However, comparative studies between paclitaxel and docetaxel are still rare, In this study, a prospective, randomized, open-label, multi-center clinical study was conducted to analyse the efficacy and safety of albumin-bound paclitaxel and docetaxel in the neoadjuvant treatment of breast cancer, and to further analyse the efficacy and safety of albumin paclitaxel in combination with chemotherapy for postoperative breast cancer in different subtypes of breast cancer patients, in order to obtain more realistic data and provide new treatment options for breast cancer patients.

DETAILED DESCRIPTION:
Neoadjuvant chemotherapy refers to systemic chemotherapy as the first step for treating breast cancer patients before planned local treatment like surgery for those without distant metastasis. It is reported that preoperative neoadjuvant chemotherapy can facilitate breast conservation, render inoperable tumors operable and provide important prognostic information at an individual patient level based on response to therapy.

Previous studies have confirmed that the efficacy of albumin-bound paclitaxel in neoadjuvant therapy and was well tolerated when combined with sequential chemotherapy with anthracyclines .

The GBG69 study was the first to compare the efficacy and safety of nab-paclitaxel (nab-P) and solvent-based paclitaxel in the neoadjuvant treatment of breast cancer. The results showed that the pCR rate in the nab-P group was significantly higher than that in the solvent paclitaxel group (38% vs 29% p<0.001). Long-term follow-up results showed that after 4 years, iDFS was also significantly improved in nab-P-treated patients compared with solvent paclitaxel (84.0% vs 76.3%; HR, 0.66; 95% CI, 0.51-0.86; P = 0.0023).

Another phase II study compared docetaxel and albumin paclitaxel in neoadjuvant chemotherapy for HER2-negative early-stage breast cancer. The results showed a slightly higher pCR rate in the nab-P group (docetaxel: 12%; nab-P: 17%). In the Ki67>20% subgroup, the pCR rates were 16% (docetaxel) vs 24% (nab-P) respectively. demonstrating that albumin-bound paclitaxel (nab-P) appears to demonstrate greater efficacy in breast cancer compared to docetaxel.

However, comparative studies between paclitaxel and docetaxel are still rare, In this study, a prospective, randomized, open-label, multi-center clinical study was conducted to analyse the efficacy and safety of albumin-bound paclitaxel and docetaxel in the neoadjuvant treatment of breast cancer, and to further analyse the efficacy and safety of albumin paclitaxel in combination with chemotherapy for postoperative breast cancer in different subtypes of breast cancer patients, in order to obtain more realistic data and provide new treatment options for breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged ≥18 years;
2. unilateral primary invasive breast cancer that meets clinical diagnostic criteria and is histologically confirmed;
3. The tumor is >2cm, and the clinical stage is consistent with cT stage 2-4; or lymph node metastasis with clear clinical/pathological evidence;
4. known hormone receptor status (estrogen receptor [ER], progesterone receptor [PR]) and HER2 status with known Ki67 expression levels; (ER/PR positive defined as stained cells >1%, HER2 positive defined as IHC 3+ or IHC 2+ with a positive FISH test);
5. Triple-negative breast cancer (TNBC): ER/PR negative, HER2 negative; tumor >2cm or lymph node metastasis with clear postoperative pathological evidence; Luminal breast cancer: ER>1%, HER2 negative, postoperative pathological evidence definite lymph node metastasis (different adjuvant chemotherapy regimens depending on whether the lymph nodes are N1 or N2-3); HER2-positive breast cancer: HER2-positive, regardless of ER/PR status; (the above classification determines enrollment and neoadjuvant therapy, and does not represent the corresponding molecular typing definition);
6. patients who need neoadjuvant chemotherapy as judged by the investigator;
7. ECOG physical fitness score of 0-1;
8. The patient has not received any treatment for breast cancer before enrollment;
9. Electrocardiogram (ECG) and echocardiography must confirm normal cardiac function within 3 months prior to randomization. Left ventricular ejection fraction (LVEF) must be ≥55%;
10. Liver and kidney function: serum creatinine ≤1.5 times the upper limit of normal; AST and ALT ≤3 times the upper limit of normal; total bilirubin ≤1.5 times the upper limit of normal, or ≤2.5 times the upper limit of normal when the patient has Gilbert's syndrome ;
11. Bone marrow function: neutrophils≥1.5×109/L, platelets≥100×109/L, hemoglobin≥90g/L;
12. Able to comply with outpatient treatment, laboratory monitoring and necessary clinical visits during the study period;
13. Subjects have the ability to understand, agree and sign the Informed Consent Form (ICF) for the study prior to initiating any protocol-related procedures; subjects have the ability to express consent (where applicable).

Exclusion Criteria:

1. Advanced and/or inoperable patients with distant metastasis confirmed by imaging evidence or pathology;
2. Patients with bilateral invasive breast cancer;
3. Other malignant tumors have occurred in the past 5 years, except for skin cancers of cured cervical carcinoma in situ and non-melanoma;
4. Pregnant or breastfeeding women; patients with childbearing potential who are unwilling or unable to take effective contraceptive measures;
5. The molecular status of ER/PR and HER2 and Ki67 cannot be determined;
6. Patients with CNS metastases or > grade 1 peripheral neuropathy;
7. Surgical axillary staging within 6 months prior to study entry;
8. Radiotherapy, chemotherapy, biotherapy and/or endocrine therapy for currently diagnosed breast cancer prior to study entry;
9. Patients with severe myelosuppression at screening;
10. Patients with severe liver dysfunction (Child's Class III) or renal dysfunction at screening ;
11. Other concomitant diseases (e.g. untreated congenital heart disease, glomerulonephritis, etc.) which, in the opinion of the investigator, seriously endanger the safety of the patient or would prevent the implementation or completion of the programme treatment;
12. Patients with hypersensitivity to any of the components of albumin paclitaxel, epirubicin, cyclophosphamide, docetaxel, trastuzumab, and pertuzumab;
13. Patients with psychiatric disorders;
14. Subjects who are participating in another clinical study or whose first dose was administered less than 4 weeks (or 5 half-lives of the study drug) from the end of the previous clinical study (last dose) ;
15. The investigator judges other situations that may affect the clinical research and the judgment of the research results and are not suitable for inclusion in the research.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1576 (Estimated)
Dates: Start 2022-07-10 (Estimated); Primary Completion 2027-06-10 (Estimated); Study Completion 2027-12-20 (Estimated)

PRIMARY OUTCOMES:
pCR(pathological complete response) | 1year
  defined as ypT0/is, ypN0 (defined as no invasive tumor in breast and axillary lymph nodes

SECONDARY OUTCOMES:
OS | 10 years
  overall survival
DFS | 2 years
  disease-free survival
DMFS | 2 years
  distant metastasis-free survival
Secondary pCR | 1 year
  defined as ypT0, ypN0 (no invasive or residual carcinoma in situ lesions in breast and axillary lymph nodes

OTHER OUTCOMES:
ORR | 1year
  tumor response rate based on imaging assessment in the neoadjuvant therapy (preoperative) stage
Remission rate of neurotoxicity | 5 years
The incidence of other AEs | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

REFERENCES:
- [Background] Robidoux A, Buzdar AU, Quinaux E, Jacobs S, Rastogi P, Fourchotte V, Younan RJ, Pajon ER, Shalaby IA, Desai AM, Fehrenbacher L, Geyer CE Jr, Mamounas EP, Wolmark N. A phase II neoadjuvant trial of sequential nanoparticle albumin-bound paclitaxel followed by 5-fluorouracil/epirubicin/cyclophosphamide in locally advanced breast cancer. Clin Breast Cancer. 2010 Feb;10(1):81-6. doi: 10.3816/CBC.2010.n.011. PMID 20133263
- [Background] Shimada H, Ueda S, Saeki T, Shigekawa T, Takeuchi H, Hirokawa E, Sugitani I, Sugiyama M, Takahashi T, Matsuura K, Yamane T, Kuji I, Hasebe T, Osaki A. Neoadjuvant triweekly nanoparticle albumin-bound paclitaxel followed by epirubicin and cyclophosphamide for Stage II/III HER2-negative breast cancer: evaluation of efficacy and safety. Jpn J Clin Oncol. 2015 Jul;45(7):642-9. doi: 10.1093/jjco/hyv055. Epub 2015 May 19. PMID 25989989
- [Background] Untch M, Jackisch C, Schneeweiss A, Conrad B, Aktas B, Denkert C, Eidtmann H, Wiebringhaus H, Kummel S, Hilfrich J, Warm M, Paepke S, Just M, Hanusch C, Hackmann J, Blohmer JU, Clemens M, Darb-Esfahani S, Schmitt WD, Dan Costa S, Gerber B, Engels K, Nekljudova V, Loibl S, von Minckwitz G; German Breast Group (GBG); Arbeitsgemeinschaft Gynakologische Onkologie-Breast (AGO-B) Investigators. Nab-paclitaxel versus solvent-based paclitaxel in neoadjuvant chemotherapy for early breast cancer (GeparSepto-GBG 69): a randomised, phase 3 trial. Lancet Oncol. 2016 Mar;17(3):345-356. doi: 10.1016/S1470-2045(15)00542-2. Epub 2016 Feb 8. PMID 26869049
- [Background] Untch M, Jackisch C, Schneeweiss A, Schmatloch S, Aktas B, Denkert C, Schem C, Wiebringhaus H, Kummel S, Warm M, Fasching PA, Just M, Hanusch C, Hackmann J, Blohmer JU, Rhiem K, Schmitt WD, Furlanetto J, Gerber B, Huober J, Nekljudova V, von Minckwitz G, Loibl S. NAB-Paclitaxel Improves Disease-Free Survival in Early Breast Cancer: GBG 69-GeparSepto. J Clin Oncol. 2019 Sep 1;37(25):2226-2234. doi: 10.1200/JCO.18.01842. Epub 2019 May 13. PMID 31082269
- [Background] Kuwayama T, Nakamura S, Hayashi N, Takano T, Tsugawa K, Sato T, Kitani A, Okuyama H, Yamauchi H. Randomized Multicenter Phase II Trial of Neoadjuvant Therapy Comparing Weekly Nab-paclitaxel Followed by FEC With Docetaxel Followed by FEC in HER2- Early-stage Breast Cancer. Clin Breast Cancer. 2018 Dec;18(6):474-480. doi: 10.1016/j.clbc.2018.06.012. Epub 2018 Jun 27. PMID 30072191